## Efficacy of Lidocaine Patch in Acute Musculoskeletal Pain in the Emergency Department: A Prospective Randomized Controlled Study.

NCT03571737

April 12, 2018

## Statistical Plan

Differences in pain scores will be analyzed using a one-tail t-test. With an a priori power analysis, we would like to see at least a 2-point difference in pain score <sup>11</sup>, with minimally clinically significant difference of 1.3 points. To achieve this, we will need at least 140 patients total (70 in each arm). Alpha will be set at 0.05, with power of 90%. Allowing for error or patient dropping out, we request that 180 people be enrolled in the study. In the study site, at least 682 patients in the month of March 2018 have come into the ED that were billed as having complaint of musculoskeletal pains.